CLINICAL TRIAL: NCT00958009
Title: A Twelve-week, Phase IIIb, Open-label, Single-arm, Multicenter Trial to Evaluate Ease of Use of a Ready-to-use, Single-use Autoinjector (SA) for Self-injection in Subjects With Relapsing Multiple Sclerosis (RMS) Treated With Rebif® 44mcg Subcutaneously (sc), Three Times a Week (Tiw)
Brief Title: The Multicenter, Open-label, Single-use Autoinjector Convenience Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: EMD Serono (Industry)
Responsible Party: Fernando Dangond, , Senior Director, Medical Affairs Neurology, EMD Serono, Inc.
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 29651
Record Dates: First submitted 2009-08-12; First posted 2009-08-13 (Estimated); Results first posted 2010-12-30 (Estimated); Last update posted 2013-08-07 (Estimated); Status verified 2013-08

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Rebidose® — The device is a ready to use single use auto injector containing Rebif® 44 mcg in a 0.5 mL prefilled syringe for sc injection

SUMMARY:
The purpose of this trial is to test the Single-Use Autoinjector for a) ease of use; b) multiple domains related to subject's acceptability and satisfaction, and c) reliability of the correct function for self-injection of Rebif® 44 mcg sc tiw in subjects with relapsing multiple sclerosis (RMS).

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects, 18-65 years of age, inclusive, at the time of informed consent signature
2. RMS diagnosed according to the McDonald criteria
3. Currently receiving Rebif® 44mcg sc tiw using manual injections and/or Rebiject II autoinjector for greater than twelve weeks
4. Capable of self-injecting using the single-use autoinjector
5. Be willing and able to comply with the study procedures for the duration of the trial
6. Have given written informed consent and signed Health Insurance Portability and Accountability Act (HIPAA) Authorization before any study-related activities are carried out
7. Female subjects must not be either pregnant or breast-feeding and must lack childbearing potential

Exclusion Criteria:

1. Have used any other injectable medications (i.e. for pain) on a regular basis during the week prior to Screening or throughout the duration of the trial (the administration of a single injection for treatment or prophylaxis of a condition unrelated to MS or Rebif® therapy (e.g., influenza or pneumococcus vaccination) will be acceptable)
2. Have received MS therapy other than Rebif® within twelve weeks prior to Screening or at any time during the trial (e.g., other disease modifying drugs, Rebif® New Formulation, combination therapy, immunomodulatory and/or immunosuppressive agents, including but not limited to any interferon, glatiramer acetate (Copolymer I), cyclophosphamide, cyclosporine, methotrexate, linomide, azathioprine, mitoxantrone, teriflunomide, laquinimod, cladribine, total lymphoid irradiation, anti-lymphocyte monoclonal antibody treatment (e.g. natalizumab, alemtuzumab/Campath, anti- CD4), Intravenous immunoglobulin (IVIg), cytokines or anti-cytokine therapy) and telbivudine
3. Have inadequate liver function, defined by a alanine aminotransferase (ALT) > 2.5x upper limit of normal (ULN), or alkaline phosphatase > 2.5x ULN, or total bilirubin > 2.5x ULN
4. Have inadequate bone marrow reserve, defined as a total white blood cell count < 3.0x 109/L, platelet count < 75x109/L, haemoglobin < 100g/L
5. Have complete transverse myelitis or bilateral optic neuritis
6. Have a history of alcohol or drug abuse
7. Have thyroid dysfunction
8. Have moderate to severe renal impairment
9. Have a major medical or psychiatric illness that in the opinion of the investigator creates undue risk to the subject or could affect compliance with the study protocol
10. Have a history of seizures not adequately controlled by treatment
11. Have serious or acute cardiac disease, such as uncontrolled dysrhythmias, uncontrolled angina pectoris, cardiomyopathy, or uncontrolled congestive heart failure
12. Have, in the opinion of the investigator, any visual, physical or cognitive impairment that would preclude the subject from self-injecting with the single-use autoinjector
13. Have a known hypersensitivity or allergy to interferon-beta or any of the excipients
14. Have participated in another clinical trial within the past thirty days
15. Are pregnant or attempting to conceive

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2009-10; Primary Completion 2010-04 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Dangond, MD, Study Director — EMD Serono
Locations (1):
- EMD Serono, Inc., Rockland, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 109 subjects were recruited from 12 US clinics in the US during the trial period Oct 2009 to April 2010.
Pre-assignment Details: Subjects who signed informed consent and satisfied the eligibility critera at screening returned to the clinic on study day 1 to begin treatment. All subjects participating in the trial received Rebif 44 mcg subcutaneious (sc, three times per week (tiw) using the single-use autoinjector (SA).
Groups:
- RMS Subject Disposition: Intent to Treat Analysis (ITT) includes all subjects who provide written informed consent and received at least one dose of trial medication
Period: Overall Study
Arm/Group | RMS Subject Disposition
Started | 109
Completed | 107
Not Completed | 2
Not completed — Adverse Event | 1
Not completed — Subject found device difficult to use | 1

BASELINE CHARACTERISTICS:
Arm/Group | RMS Subject Disposition
Number analyzed (Participants) | 109
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 109
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 46.0 (9.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 76
  Male | 33
Region of Enrollment [Number; unit: participants]
  United States | 109

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Relapsing Multiple Sclerosis (RMS) Subjects Rating the Single-use Autoinjector as 'Easy to Use' or 'Very Easy to Use' for Self-injection in a User Trial Questionnaire
Description: Data from the User Trial Questionnaire, Question 14 (Overall, how do you rate your experience with using the injection device?) Mean and confidence interval refer to proportion of subjects responding positively to question. Missing values were replaced with worst case response.
Time Frame: at 12 weeks
Population: Subjects in the all enrolled analysis set who received at least one dose of investigational medicinal product (IMP) were included in the ITT analysis set. This analysis set was used to analyze the primary and secondary variables and all safety data.
Measure: Mean (95% Confidence Interval); unit: Proportion of subjects
Arm/Group | RMS Subject Disposition
Number analyzed (Participants) | 109
Proportion of subjects | 0.86 [0.80 to 0.93]
Statistical Analysis 1: Comparison: RMS Subject Disposition; Test type: Superiority or Other; mean positive response = 0.86, 95% CI 2-sided [0.80 to 0.93] — Confidence Interval calculated from normal approximation to the binomial. The primary objective was met if the lower bound of the 95% confidence interval is >0.50

2. Secondary Outcome: Multiple Secondary Endpoints Were Assessed, Based on Questions From the User Trial Questionnaire Related to the Single-use Autoinjector Device Use-related Outcomes.
Description: The User Trial Questionnaire was used to assess the ease of use, functional reliability, overall satisfaction with device attributes, convenience, safety and portability of the device. Mean and confidence intervals refer to proportion of subjects responding positively to question. Secondary endpoints presented for decriptive purposes only thus no statistical analysis performed.
Time Frame: at 12 weeks
Population: Subjects in the all enrolled analysis set who received at least one dose of IMP were included in the ITT analysis set. This analysis set was used to analyze the primary and secondary variables and all safety data.
Measure: Mean (95% Confidence Interval); unit: Proportion of subjects
Arm/Group | RMS Subject Disposition
Number analyzed (Participants) | 109
Proportion of subjects
  Device makes injections simple | 0.83 [0.77 to 0.90]
  Allows easy access to skin injection sites | 0.78 [0.70 to 0.86]
  Helps me self-administer injections | 0.83 [0.75 to 0.90]
  Ease of pushing device against skin | 0.76 [0.68 to 0.84]
  Ease of holding device during injection | 0.77 [0.69 to 0.85]
  Able to often or always administer full injection | 0.96 [0.93 to 1.00]
  Satisfaction with size of device | 0.61 [0.51 to 0.70]
  Satisfaction with ease of removing cap from device | 0.87 [0.81 to 0.93]
  Satisfaction with ease of activating button | 0.78 [0.70 to 0.86]
  Satisfaction with time to inject medicine | 0.83 [0.75 to 0.90]
  Satisfaction with ability to see post injection | 0.81 [0.73 to 0.88]
  Rate convenience of device | 0.74 [0.66 to 0.83]
  Rate how reliable injection device was | 0.79 [0.71 to 0.87]

ADVERSE EVENTS:
Arm/Group | RMS Subject Disposition
Serious Adverse Events (participants affected / at risk) | 4/109
Other Adverse Events (participants affected / at risk) | 83/109
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RMS Subject Disposition (N=109)
Chest Pain (General disorders) | 1 (1)
Angina pectoris (Cardiac disorders) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1)
Convulsion (Nervous system disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RMS Subject Disposition (N=109)
Influenza like illness (General disorders) | 26 (26)
Injection site erythema (General disorders) | 39 (39)
Injection site haematoma (General disorders) | 13 (13)
Injection site pain (General disorders) | 27 (27)
Injection site swelling (General disorders) | 8 (8)
Upper respiratory tract infection (Infections and infestations) | 6 (6)
Headache (Nervous system disorders) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Neither Institution nor any Principal Investigators shall publish or present any results from such Study to any third parties until: (i) EMD Serono publishes the results from all sites participating in such Study; (ii) Institution receives notification from EMD Serono that publication of the multi-site results is no longer planned; or (iii) twenty-four (24) months following the completion of the multi-site study at all sites, whichever occurs first.